CLINICAL TRIAL: NCT00558740
Title: Effects of Dietary Proteins on Hepatic Lipid Metabolism
Status: Completed | Type: Observational
Sponsor: University of Lausanne (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Prof. L uc Tappy, Department of Physiology, University of Lausanne
Other Study IDs: protocol 66/07/CE/FBM; SNF 310000-109737
Record Dates: First submitted 2007-11-14; First posted 2007-11-15 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2009-11

CONDITIONS: Metabolic Syndrome X
Keywords: Dietary protein; Fructose; VLDL-triglycerides; Hepatic de novo lipogenesis; Lipid oxidation
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- healthy volunteers
  Interventions: Other: high protein intake

INTERVENTIONS:
Other: high protein intake — acute high protein intake chronic (6-day) high protein intake acute+chronic high protein intake control

SUMMARY:
Individuals submitted to a high-fat or a high-fructose/sucrose diet develop, over a 6 day-period, several features of the metabolic syndrome, including increased plasma triglycerides, increased intrahepatic lipids, and decreased hepatic insulin sensitivity. It has been recently observed that the increase in intrahepatic lipids observed after a high fat diet is largely prevented when protein intake is concomitantly increased. This suggests that dietary protein protects the liver against some of the deleterious effects of a high fat diet. Mechanisms underlying this effect of protein may include an increased hepatic fat oxidation.

The aims of this study are:

1. to evaluate the effects of dietary protein on several major pathways involved in hepatic lipid metabolism ( ketogenesis, lipid oxidation, de novo lipogenesis, VLDL-triglyceride secretion
2. to determine whether the decrease in intra-hepatic lipids observed when dietary protein intake is increased are to be attributed to acute or long-term effects of proteins

DETAILED DESCRIPTION:
This research project include three sub-studies of healthy, normal weight, young males.

Sub-study A1: The effects of acute and chronic increase in protein intake on whole body and hepatic lipid metabolism will be studied in healthy males. Two groups of 7 subjects will be recruited.

One group will be studied on three occasions, during which their metabolism will be evaluated in basal, post-absorptive conditions and over 6 hours after ingestion of mixed meal containing carbohydrate, fat (including medium chain triglycerides (MCT) labeled with 13C3 tri-octanoate), and protein.

* control: on one occasion subjects will have received an isocaloric diet (55% carbohydrate, 30% fat, 15% protein) during 4 days. On the morning of the 5th day, they will be studied for 2 hours in basal, postabsorptive conditions and over 6 hours following ingestion of a meal providing ca 10 kcal /kg body weight and containing 55% carbohydrate, 35% fat (of which 15% medium chain triglycerides (MCT) labeled with 13C3 trioctanoate, and 10% protein.
* acute increase in protein intake: on the second occasion, they will have received an isocaloric diet (55% carbohydrate, 30% fat, 15% protein) during 4 days. On the morning of the 5th day, they will be studied for 2 hours in basal, post absorptive conditions and over 6 hours following ingestion of a meal providing ca 12.5 kcal /kg body weight and containing 45% carbohydrate, 30% fat (of which 13% medium chain triglycerides (MCT) labeled with 13C3 trioctanoate, and 25% protein.
* chronic high protein intake: on the third occasion, they will have received an hypercaloric diet ( 130% energy requirement, providing 42% carbohydrate, 23% fat, 35% protein; this corresponds to the isocaloric diet given on the first two occasions, additioned with 1g/day protein) during 4 days. On the morning of the 5th day, they will be studied for 2 hours in basal, post absorptive conditions and over 6 hours following ingestion of a meal providing ca 12.5 kcal /kg body weight and containing 45% carbohydrate, 30% fat (of which 13% medium chain triglycerides (MCT) labeled with 13C3 trioctanoate) and 25% protein. The three tests will be done in a randomized order, with a washout period of at least 4 weeks between each test.

On each occasion, the following parameters will be monitored in basal conditions and after ingestion of the mixed meal.

Deuterated glucose (6,6 2H2-glucose) and glycerol (2H5 glycerol) will be infused throughout the tests. Measurements will be include:

* whole body energy expenditure and net substrate oxidation (indirect calorimetry)
* plasma glucose, free fatty acids, VLDL-TG, ketone bodies, insulin, glucagon, growth hormone
* MCT oxidation (breath 13CO2)
* Glucose and glycerol turnover
* VLDL kinetics (modelization of 2H5 incorporation into VLDL-triglycerides. Sub-study A2: A second group of 7 subjects will be studied on three occasions according to the same protocol, except that the test meal will not include MCT and that long-chain triglycerides (LCT) will be labeled with 13C3 triolein. The same metabolic parameters will be recorded, except for MCT oxidation, which will be replaced by LCT oxidation.

This sub-study will allow to evaluate the hypothesis that dietary proteins enhance whole body hepatic lipid oxidation and decrease hepatic VLDL-triglyceride secretion.

Sub-study B: The effects of acute and chronic increase in protein intake on fructose-induced hepatic de-novo lipogenesis and VLDL-triglyceride secretion will be studied in healthy males. One group of 8 subjects will be recruited.Each subject will be studied on 4 separate occasions during which their metabolism will be studied for 2 hours in basal conditions and over 6 hours after ingestion of a standard test meal containing 0.75 g/kg fructose labeled with 13C6 fructose and 0.3 or 0.8 g/kg protein.

* control: subjects will be studied after 6 days of a a high fructose diet (isocaloric diet containing 45 % complex carbohydrate, 10% sugars, 30% fat, and 15% protein, additionned with 3.0 g/kg body weight/day fructose) and measurements will be performed in basal conditions and after administration of a standard test meal with 0.3 g/kg protein.
* acute effects of protein: subjects will be studied after 6 days of a high fructose diet, and measurements will be performed in basal conditions and after administration of a standard test meal with 0.8 g/kg protein
* Chronic effects of high protein: subjects will be studied after 6 days of a high fructose diet additionned with 1g/kg body weight protein/day and after administration of a standard test meal with 0.3 g/kg protein.
* Chronic + acute effects of high protein: subjects will be studied after 6 days of a high fructose diet additionned with 1g/kg body weight protein/day and after administration of a standard test meal with 0.8 g/kg protein

Deuterated glucose (6,6 2H2 Glucose) and glycerol (2H5 glycerol) will be infused throughout the tests. Measurements will be include:

* whole body energy expenditure and net substrate oxidation (indirect calorimetry)
* plasma glucose, free fatty acids, VLDL-TG, ketone bodies, insulin, glucagon, growth hormone
* Fructose oxidation (breath 13CO2)
* Hepatic de novo lipogenesis (13C VLDL-palmitate)
* Gluconeogenesis (13C glucose)
* Glucose and glycerol turnover
* VLDL kinetics (modelization of 2H5 incorporation into VLDL-triglycerides This sub-study will allow to evaluate the hypothesis that dietary proteins inhibit hepatic de-novo lipogenesis and enhance the oxidation of fructose.

Subcutaneous adipose tissue biopsies will be obtained on two occasions, ie after high protein and control diet for analysis of gene expression.

Sub-study B3:The effects of hyperglucagonemia on fructose-induced hepatic de-novo lipogenesis and VLDL-triglyceride secretion will be studied in healthy males. One group of 6 subjects will be recruited.Each subject will be studied on 2 separate occasions during which their metabolism will be studied for 2 hours in basal conditions and over 8 hours after ingestion of a standard test meal containing 0.75 g/kg fructose labeled with 13C6 fructose and 0.3 g/kg protein.

* control: subjects will be studied after 6 days of an energy balanced diet and measurements will be performed in basal conditions and after administration of a standard test meal with 0.75g/g 13C-labelled fructose and 0.3 g/kg protein.
* acute effects of glucagon: subjects will be studied after 6 days of an energy balanced diet and measurements will be performed in basal conditions and after administration of a standard test meal with 0.75g/g 13C-labelled fructose and 0.3 g/kg protein together with a glucagon infusion (5ng/kg/min)

Deuterated glucose (6,6 2H2 Glucose) and glycerol (2H5 glycerol) will be infused throughout the tests. Measurements will include:

* whole body energy expenditure and net substrate oxidation (indirect calorimetry)
* plasma glucose, free fatty acids, VLDL-TG, ketone bodies, insulin, glucagon, growth hormone
* Fructose oxidation (breath 13CO2)
* Hepatic de novo lipogenesis (13C VLDL-palmitate)
* Gluconeogenesis (13C glucose)
* Glucose and glycerol turnover
* VLDL kinetics (modelization of 2H5 incorporation into VLDL-triglycerides This sub-study will allow to evaluate the hypothesis that dietary proteins inhibit hepatic de-novo lipogenesis and enhance the oxidation of fructose.

through an increased glucagon secretion

ELIGIBILITY:
Inclusion Criteria:

* age 18-30
* sex male
* BMI 19-25 kg/m2
* sedentary
* good physical health

Exclusion Criteria:

* family history of diabetes
* use of drugs or illicit substances
* consumption of alcohol >50 g/week
* vegetarians
* smokers

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Whole body lipid oxidation Medium chain triglyceride oxidation Long chain triglyceride oxidation VLDL-triglyceride kinetics Hepatic de novo lipogenesis whole body glucose and glycerol turnover | acute effects of dietary proteins and after 4 days on a high protein day

SECONDARY OUTCOMES:
Energy expenditure Glucagon/insulin ratio Plasma growth hormone concentrations gene expression in subcutaneous adipose tissue Plasma ketone bodies concentrations | acute effects of dietary proteins and after 4 days on a high protein day

CONTACTS AND LOCATIONS:
Overall Officials: l Tappy, MD, Principal Investigator — University of Lausanne
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland